CLINICAL TRIAL: NCT00511628
Title: BMI-2002 Study: Evaluation of Functionality and Evolution of Body Weight of Psychotic Patients With a High Body Mass Index
Brief Title: Study on the Safety of Risperidone on Obese or Overweight Patients With Schizophrenia
Status: Terminated | Type: Observational
Why Stopped: Due to the achievement of minimum required sample size and new changes in local regulations.
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Country Medical Director, Janssen-Cilag S.A., Spain
Other Study IDs: CR009313
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Risperidone; Schizoaffective disorder; Schizophreniform disorder; Weight gain
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Weight Gain | interventions — Risperidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001: Risperidone As prescribed
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — As prescribed

SUMMARY:
The purpose of this study is to evaluate the safety of risperidone treatment in patients who are overweight and/or obese.

DETAILED DESCRIPTION:
This is an observational, multicenter, open and prospective study. The primary objective is to evaluate safety of risperidone in patients who are overweight and/or obese. It is expected to enroll 1500 patients with Schizophrenia or Schizoaffective disorder, in which physicians considered the use of risperidone as treatment under clinical practice with a BMI (Body Mass Index) >25, or for patients that have increased their body weight >7% in the last year with the previous treatment (even with a BMI< 25), and for patients that have shown intolerance to a previous antipsychotic treatment. The study drug is risperidone, 3-6 mg per day, orally, during the study period (6 months). All data collected will be prospective and will include the following: demographic data, psychiatric history and comorbidities, concomitant treatment, body weight, treatment history , other illness related to obesity ( such as diabetes mellitus I & II, hypertension and hypercholesterolemia) and adverse events. Observational Study: Risperidone, 3-6 mg per day, orally, during the study period (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Schizophrenia or Schizoaffective disorder, in which physicians considered the use of risperidone as treatment under clinical practice with a BMI >25
* Patients have increased their body weight >7% in the last year with the previous treatment even with a BMI< 25
* Patients that have shown intolerance to a previous antipsychotic treatment

Exclusion Criteria:

* Pregnant or lactating patients
* Patients with psychiatry pathology other than Schizophrenia or schizoaffective disorder
* Patients with neurology pathology except Parkinsonism induced by neuroleptics
* Patients with other severe concomitant pathology
* Patients treated with Risperidone in the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Schizophrenia or Schizoaffective disorder, in which physicians considered the use of risperidone as treatment under clinical practice with a BMI >25; Patients have increased their body weight >7% in the last year with the previous treatment even with a BMI< 25 ; Patients that have shown intolerance to a previous antipsychotic treatment
Sampling Method: Non-Probability Sample
Enrollment: 1717 (Actual)
Dates: Start 2001-07; Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation of Risperidone in patients who are overweight and/or obese | 6 months

SECONDARY OUTCOMES:
Effectiveness | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.

REFERENCES:
- See also: Study on the safety of risperidone on obese or overweight patients with schizophrenia. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=284&filename=CR009313_CSR.pdf